CLINICAL TRIAL: NCT06352346
Title: Evaluation of a Compensatory Brain Game Supporting Goal Management Training Intervention Targeting Executive Function in Acquired Brain Injury Patients With Depressive and/or Anxiety Symptoms: a Single-case Experimental Design
Brief Title: A Single-case Design to Investigate a Compensatory Brain Game Supporting Goal Management Training Intervention in a Psychiatric Brain Injury Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProPersona (Other)
Responsible Party: Principal Investigator, Helen Alexandra Anema, Principal Investigator, ProPersona
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Plan Game_ABI&Psychiatry
Record Dates: First submitted 2024-03-29; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Acquired Brain Injury; Depressive Symptoms; Anxiety; Executive Dysfunction
Keywords: Goal Management Training; Compensatory Strategy Training; Serious Gaming
MeSH Terms: conditions — Brain Injuries; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A randomized Single-case Experimental Design (SCED) with a follow-up period of 6 weeks. Participants will be first assigned to a baseline phase (phase A). The start of the treatment phase (phase B) is determined randomly for each participant, given the restriction that the baseline phase (phase A) should last for at least three weeks (21 days) and at most five weeks (30 days). This means that the treatment phase can start on any day between the 21th and the 30th days. So, in the first three weeks, all participants are in the baseline condition. The duration of baseline will thus be different for each subject. Nonspecific effects, such as linear trends, retesting or non-specific recovery, can be controlled by this approach, since expected changes in level of performance due to treatment should parallel this stepwise onset of therapy procedure.
  Phase A acts as a control and is therefore compared with phase B.
Who Masked: Outcomes Assessor
Masking Description: The target behavior (i.e. performance on an untrained shopping task) will be measured repeatedly, on a minimum of six occasions in each phase where possible, in accordance with the recommendations of the What Works Clearinghouse and RoBiNT criteria. Repeated measures of target behavior will be assessed via the OxMET-NL task and is scored automatically: no assessor input is required to either save or score the main outcome data. The secondary outcome measure(s) are scored by an outcome assessor who is blind to the order in which the secondary outcome measure(s) were taken.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Intervention: Baseline phase (Phase A) (No Intervention): o At the start of the study, all participants are assigned to the baseline phase (phase A). During phase A, patients do not receive interventions related to executive function problems. The start of the intervention phase (phase B) is determined randomly for each participant, given the restriction that phase A should last for at least three weeks (21 days) and at most five weeks (30 days). This means that phase B can start on any day between the 21th and the 30th days, resulting in a total of 10 possible assignments. So, in the first three weeks, all participants are in phase A. The duration of phase A will thus be different for each subject. Phase A acts as a control and is therefore compared with phase B.
- Experimental: Intervention phase (Phase B): Goal Management Training (Experimental): During the intervention phase (phase B), all included participants will have 6 sessions of Goal Management Training (GMT; twice per week) in which two individual chosen IADL-tasks will be subdivided into multiple steps under guidance of a therapist using the GMT method. In addition participants play the compensatory brain game in which they are challenged to apply the learned GMT strategy in an imaginary and safe environment.
  Interventions: Behavioral: Compensatory brain game supporting Goal Management Training intervention
- Follow-up period (No Intervention): A follow-up period of six weeks takes place after phase B. During this follow-up period, patients receive no intervention.

INTERVENTIONS:
Behavioral: Compensatory brain game supporting Goal Management Training intervention — o The investigational treatment is only given during the intervention phase (phase B), and consists of six treatment sessions. In the treatment sessions, patients learn and apply the GMT algorithm. This means that the multiple steps of the GMT as well as the actual performance of the IADL-task goals will be learned under guidance of a therapist. In order to facilitate generalization, patients will learn to use the algorithm during the performance of untrained tasks by playing the treatment supporting Plan Game. Because of this, patients are able to practice the application of the GMT algorithm independently outside the therapy session. Besides, the intervention also includes a Plan Tool. This is a mobile application that can be used as an aid during the performance of (instrumental) activities of daily living (IADL) tasks in order to perform activities more independently. The GMT treatment sessions are given twice a week (max. 60 minutes for each attendance).
  Arms: Experimental: Intervention phase (Phase B): Goal Management Training

SUMMARY:
The main cognitive complaint in brain-injured patients is often the everyday disorganization caused by Executive Function (EF) deficits. EF deficits are often seen in patients with psychiatric disorders i.e. depression or anxiety. In order to minimize everyday disorganization, effective EF interventions are required. Interventions using compensatory strategies have the potential to enable patients to minimize disabilities, minimize participation problems and to function more independently in daily life. A well-known evidence-based intervention that uses compensatory strategies is Goal Management Training (GMT), a training that has been found to alleviate depressive symptoms in a depressed population. GMT entails learning and applying an algorithm, in which a daily task is subdivided into multiple steps to handle executive difficulties of planning, and problem solving. To adopt the GMT strategy and ensure maximal profitability for patients, they have to learn to use the algorithm in different situations and tasks. Therefore, GMT is comprehensive, time-consuming and thus labour-intensive. Along with this, brain games become increasingly attractive as an (add-on) intervention, most notably in an effort to develop home-based personalized care. Until now, however, the rationale behind brain games is based on what can be considered the restorative approach (i.e. strengthening of executive problems) rather than practicing compensatory strategies, with little or no transfer to improvements in daily life functioning. This study therefore aims to assess the potential of a newly developed Brain Game, based on compensatory strategies, as an add-on to GMT to develop a shortened and partly self-paced GMT intervention. The primary objective of this study is to assess whether the use of a compensatory brain game supported GMT treatment could be of interest in people with EF deficits after ABI that also suffer from depression or anxiety, to improve goal achievement, their executive function performance during goal-related tasks, and their executive performance during an ecological valid shopping task. Also we assess whether psychological symptoms alleviate following the GMT intervention and at 6-weeks follow-up. The study will be a multiple-baseline across individuals single-case experimental design (SCED). The study population consists of brain-injured patients, between 18 and 75 years old that receive in-patient mental neuropsychiatric healthcare. Participants eligible for the study must have EF deficits due to (nonprogressive) Acquired Brain Injury (ABI), minumum time post-onset of 3 months and depressive or anxiety symptoms. EF deficits will be assessed by extensive neuropsychological examination. Participants will be recruited from an inpatient clinic. In the course of one and a half year four participants will be recruited.

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 75 years
* Non-progressive acquired brain injury
* Minimal time post-onset of 3 months
* Receive inpatient neuropsychiatric care at the time of inclusion
* Executive deficits (neuropsychological assessment)
* Reasonable amount of awareness in their deficits, at least to the extent that they are motivated and capable to learn new skills with respect to their executive performance.

Exclusion Criteria:

* Inability to speak/understand the Dutch language
* Severe psychiatric disorders such as psychosis, manic episode, severe disruptive behavior
* Neurodegenerative disorders (i.e. dementia, Huntington, Parkinson
* Substance abuse (active)
* Severe cognitive comorbidity (i.e. Korsakov)
* Aphasia
* Neglect
* Unable to look at a computer screen for 15 minutes
* Unable to operate a keyboard or computer mouse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in performance on the Oxford Multiple Errands Test- Dutch version (OxMET-NL) from phase A to phase B | The target behavior (i.e. performance on the OxMET-NL) will be measured repeatedly, two times a week, for the duration of phase A (3 to 5 weeks) and phase B (36 weeks
  The target behavior will be assessed repeatedly, on a minimum of six occasions in phase A and B, in accordance with the recommendations of the What Works Clearinghouse and RoBiNT criteria (Tate et al., 2013). The OxMET-NL task is a computer-tablet based version of the Multiple Errands Test and is scored automatically. The task requires patients to buy six items and to answer two questions. The main outcome measure of the task is accuracy which ranges from -10 to + 10 (higher score is better outcome) based on a score obtained in each shop.

SECONDARY OUTCOMES:
Change on the Visual Analogue Scale (VAS) from phase A to phase B to follow-up | The VAS will be assessed repeatedly, two times a week, for the duration of phase A (3 to 5 weeks), phase B (3 weeks) and follow-up (6 weeks)
  Subjective experience of strategy use in daily life and during the performance of instrumental activities of daily living (IADL) and three psychological symptoms. Scale ranges from 0-100 of which higher scores means better outcome.
Change in performance on treatment goals as measured with the Goal Attainment Scale (GAS) | pre-intervention, immediately following intervention and at six weeks follow-up
  GAS is a mathematical technique for quantifying the achievement of goals set, used in rehabilitation. GAS is described as a method of scoring the extent to which patient's individual goals are achieved in the course of intervention. In effect, each patient has his or her own outcome measure, but this is scored in a standardized way as to allow statistical analysis. The achievement of each goal (IADL-task) can be measured on a 5-point scale ranging from -2 to +2. Outcomes can be quantified in a single aggregated goal attainment score. This method gives a numerical T-score which is normally distributed about a mean of 50 (if the goals are achieved precisely) with a standard deviation of around this mean of 10 (if the goals are overachieved or underachieved).
Change in performance on two trained IADL task (treatment goals) | pre-intervention, immediately following intervention and at six weeks follow-up
  Performance on two treatment goals is measured with a standardised scale . The tasks will be divided into multiple steps using the GMT method. Each task step will be assessed following a 3-point scale (ranging from 2=competent to 0=deficit). Total scores per task will be adjusted to a 100-point scale using the following formula: performance = (total score / (number of steps × 2)) × 100. Thus, a performance of 100% indicating perfect IADL task performance.
Change in everyday difficulties in activities/participation as measured on the Daily Living Questionnaire (DLQ-R-NL) | pre-intervention, immediately following intervention and at six weeks follow-up
  The Dutch version of the Daily Living Questionnaire measures how much mental or cognitive difficulty the participant generally has by performing daily activities. Scale ranges from 0-112 of which higher scores means better outcome.
Change in strategy use during the performance of trained and untrained IADL tasks | pre-intervention, immediately following intervention and at six weeks follow-up
  A self-designed questionnaire to examine self-reported strategy use will also be administered after the performance of the trained and untrained IADL tasks in order to measure strategy use in a traditional memory task. First, participants are openly asked which strategies they use during the performance of an IADL task. Subsequently, they are given a list with possible strategy components of GMT that one could use to perform a task and are asked to place a check mark next to each strategy that they had used.
Change in subjective experience of strategy use in daily life | pre-intervention, immediately following intervention and at six weeks follow-up
  GMT strategy use is assessed through an adjustment of the Strategy Use Inventory; SUI . Participants have to indicate how often they use a certain strategy in daily life situations using a 5-point rating scale ranging from 1 (never) to 5 (often) which implies that higher scores mean better outcome. Average item scores are calculated
Change in subjectively experienced psychological symptoms such as depressive, anxiety and stress symptoms. | pre-intervention, immediately following intervention and at six weeks follow-up
  Psychological symptoms are measured with the DASS-42. The DASS is a 42-item self-report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress on a 4-point rating scale Subscale scores are calculated by summarizing the item scores, ranging from 0-42. A higher score means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- ProPersona, Wolfheze, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tate RL, Perdices M, Rosenkoetter U, Wakim D, Godbee K, Togher L, McDonald S. Revision of a method quality rating scale for single-case experimental designs and n-of-1 trials: the 15-item Risk of Bias in N-of-1 Trials (RoBiNT) Scale. Neuropsychol Rehabil. 2013;23(5):619-38. doi: 10.1080/09602011.2013.824383. Epub 2013 Sep 9. PMID 24050810
- [Background] Bertens D, Kessels RP, Boelen DH, Fasotti L. Transfer effects of errorless Goal Management Training on cognitive function and quality of life in brain-injured persons. NeuroRehabilitation. 2016;38(1):79-84. doi: 10.3233/NRE-151298. PMID 26889801
- [Background] Dechamps A, Fasotti L, Jungheim J, Leone E, Dood E, Allioux A, Robert PH, Gervais X, Maubourguet N, Olde Rikkert MG, Kessels RP. Effects of different learning methods for instrumental activities of daily living in patients with Alzheimer's dementia: a pilot study. Am J Alzheimers Dis Other Demen. 2011 Jun;26(4):273-81. doi: 10.1177/1533317511404394. Epub 2011 Apr 17. PMID 21502092
- [Background] Frankenmolen NL, Overdorp EJ, Fasotti L, Claassen JAHR, Kessels RPC, Oosterman JM. Memory Strategy Training in Older Adults with Subjective Memory Complaints: A Randomized Controlled Trial. J Int Neuropsychol Soc. 2018 Nov;24(10):1110-1120. doi: 10.1017/S1355617718000619. Epub 2018 Aug 31. PMID 30168408
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811